CLINICAL TRIAL: NCT06445452
Title: The Impact of SNAP-Ed on Dietary Quality, Food Safety Handling Behaviors, and Insulin Resistance Among Bhutanese Adults Residing in New Hampshire
Brief Title: The Impact of SNAP-Ed Among Bhutanese Adults Residing in New Hampshire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Responsible Party: Principal Investigator, Sherman Bigornia, Assistant Professor, University of New Hampshire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNH-13-FY2022_38-01
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Supplemental Nutrition Assistance Program Education; Bhutanese Refugee Adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAP-Ed (Experimental)
  Interventions: Behavioral: Direct SNAP-Ed
- No SNAP-Ed (Placebo Comparator)
  Interventions: Behavioral: Direct SNAP-Ed

INTERVENTIONS:
Behavioral: Direct SNAP-Ed — Six in-home SNAP-Ed lessons are delivered to participants in the SNAP-Ed arm. Lessons are offered weekly and directed by a bilingual and bicultural community health worker.

SUMMARY:
The goal of this pilot randomized controlled trial is to test the potential efficacy of Supplemental Nutrition Assistance Program Education (SNAP-Ed) among Bhutanese refugee adults residing in New Hampshire. The main questions are whether direct SNAP-Ed delivered through 6 lessons affects dietary quality and biomarkers of metabolic risk. Participants in the SNAP-Ed arm will be asked to participate in weekly lessons delivered in their homes by a bicultural and bilingual nutrition educator. Individuals in the control group did not receive SNAP-ED. All participants will be asked to complete surveys and provide blood and fecal samples prior at baseline and at the end of the study period (7 to 8 weeks).

ELIGIBILITY:
Inclusion criteria are (1) identifies as a Bhutanese refugee (2) 18 years and older (3) does most of the cooking and shopping for his/her household. Exclusion Criteria are (1) has been told by her/his doctor that she/he has diabetes (2) history of use of glucose lowering medications (3) pregnant or trying to become pregnant (4) currently diets for weight loss or dietary restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Index Score | 0 and 7-8 weeks
  All participants will provide three 24-hr recalls at baseline and the exit visit. Dietary intake will be average across the three recalls. The HEI score rubric will be applied to the dietary intakes where a higher score indicates greater adherence to the US Dietary Guidelines.
Glucose Homeostasis Biomarkers | 0 and 7-8 weeks
  Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) is calculated using fasting insulin and glucose values, where a higher values indicates greater insulin resistance. HbA1c will also be measured.
Lipid Panel | 0 and 7-8 weeks
  Total cholesterol, LDL-Cholesterol, HDL-Cholesterol and triglycerides will be measured as an indicators of CVD risk.
Inflammatory Biomarkers | 0 and 7-8 weeks
  TNF-alpha, C-Reactive Protein, and IL-6 will be measured where higher values indicate greater inflammation.
Gut Microbiome Composition | 0 and 7-8 weeks
  Outcomes include short-chain fatty acids (Akkermansia municiphilla, Ruminococcus bromii, Faecalibacterium prausnitzii, Eubacterium rectale, and Eubacterium hallii) and lower abundance of those that synthesize branched-chain amino acids (Bacillus-Lactobacillus-Streptococcus groups, and Proteobacteria). In addition, gut microbial diversity will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Building Community in New Hampshire, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No